CLINICAL TRIAL: NCT00237809
Title: D-Serine Treatment of Negative Symptoms and Cognitive Deficits in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Donaghue Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Deepak C. D'Souza, Associate Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23594; DF01-015
Record Dates: First submitted 2005-09-13; First posted 2005-10-12 (Estimated); Results first posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Drug and control CRT (Experimental): D-serine/control
  Interventions: Drug: D-serine; Behavioral: Cognitive Retraining Placebo
- Drug and CRT (Experimental): D-serine/cog rehab
  Interventions: Drug: D-serine; Behavioral: Cognitive Retraining (CRT)
- Placebo Drug and Placebo CRT (Experimental): Placebo/control
  Interventions: Drug: Placebo; Behavioral: Cognitive Retraining Placebo
- Placebo Drug and CRT (Experimental): Placebo/cog rehab
  Interventions: Behavioral: Cognitive Retraining (CRT); Drug: Placebo

INTERVENTIONS:
Drug: D-serine — D-serine (30 mg/kg)
  Arms: Drug and CRT; Drug and control CRT
Behavioral: Cognitive Retraining (CRT) — Cognitive retraining therapy (CRT)
  Arms: Drug and CRT; Placebo Drug and CRT
Drug: Placebo — Placebo D-serine Drug
  Arms: Placebo Drug and CRT; Placebo Drug and Placebo CRT
Behavioral: Cognitive Retraining Placebo — Cognitive retraining therapy (CRT) control
  Arms: Drug and control CRT; Placebo Drug and Placebo CRT

SUMMARY:
This study is based on the hypothesis that by increasing N-methyl-D-aspartic acid (NMDA) receptor function in the brain and thereby increasing the capacity of the brain to both form new connections and strengthen existing connections, schizophrenic patients may derive both greater and sustained benefit from cognitive retraining.

DETAILED DESCRIPTION:
Patients with schizophrenia or schizoaffective disorder who are currently receiving antipsychotic medication will be randomly assigned in a double-blind manner to receive either D-serine (30 mg/kg) or placebo in addition to cognitive rehabilitation or a non-interactive placebo for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder

Exclusion

* Pregnant or lactating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2002-09; Primary Completion 2010-12 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak C D'Souza, M.D., Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Connecticut Mental Health Center, New Haven, Connecticut
  - VA Connecticut Healthcare System, West Haven, Connecticut

REFERENCES:
- [Background] Tsai GE, Yang P, Chung LC, Tsai IC, Tsai CW, Coyle JT. D-serine added to clozapine for the treatment of schizophrenia. Am J Psychiatry. 1999 Nov;156(11):1822-5. doi: 10.1176/ajp.156.11.1822. PMID 10553752
- [Background] Tsai G, Yang P, Chung LC, Lange N, Coyle JT. D-serine added to antipsychotics for the treatment of schizophrenia. Biol Psychiatry. 1998 Dec 1;44(11):1081-9. doi: 10.1016/s0006-3223(98)00279-0. PMID 9836012
- [Background] Heresco-Levy U, Javitt DC, Ebstein R, Vass A, Lichtenberg P, Bar G, Catinari S, Ermilov M. D-serine efficacy as add-on pharmacotherapy to risperidone and olanzapine for treatment-refractory schizophrenia. Biol Psychiatry. 2005 Mar 15;57(6):577-85. doi: 10.1016/j.biopsych.2004.12.037. PMID 15780844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between 2003 and 2008, with enrollment of subjects in India starting later (2005) and ending in 2008.
Pre-assignment Details: 132 subjects were screened for eligibility. After screening, eligible subjects were randomized to receive: D-serine+CRT, placebo D-serine+CRT, D-serine + control CRT, or placebo D-serine + control CRT. Randomization was stratified by screening performance IQ. Separate randomization schedules (block size= 4) were generated within IQ stratum.
Groups:
- D-serine Drug /CRT Placebo: D-serine/control
  D-serine : D-serine (30 mg/kg)
- Placebo Drug /CRT: Placebo/cog rehab
  Cognitive retraining : Cog rehab
- D-serine Drug/CRT: D-serine/cog rehab
  D-serine : D-serine (30 mg/kg)
- Placebo Drug/ Placebo CRT: Placebo/control
Period: Overall Study
Arm/Group | D-serine Drug /CRT Placebo | Placebo Drug /CRT | D-serine Drug/CRT | Placebo Drug/ Placebo CRT
Started | 27 | 27 | 24 | 26
Completed | 16 | 17 | 15 | 17
Not Completed | 11 | 10 | 9 | 9
Not completed — Lost to Follow-up | 11 | 10 | 9 | 9

BASELINE CHARACTERISTICS:
Groups:
- D-serine/Control: D-serine/control
  D-serine : D-serine (30 mg/kg)
- Placebo/Cog Rehab: Placebo/cog rehab
  Cognitive retraining : Cog rehab
- D-serine/Cog Rehab: D-serine/cog rehab
  D-serine : D-serine (30 mg/kg)
- Placebo/Control: Placebo/control
  Cognitive retraining : Cog rehab
- Total: Total of all reporting groups
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control | Total
Number analyzed (Participants) | 27 | 27 | 24 | 26 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7500 (8.01889) | 34.4762 (8.76139) | 36.3158 (9.16547) | 34.4545 (9.36420) | 35.21 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 5 | 7 | 26
  Male | 18 | 22 | 19 | 19 | 78

OUTCOME MEASURES:

1. Primary Outcome: Wisconsin Card Sorting Test (WCST)
Description: The WCST allows the clinician to speculate to the following "frontal" lobe functions: strategic planning, organized searching, utilizing environmental feedback to shift cognitive sets, directing behavior toward achieving a goal, and modulating impulsive responding. The test can be administered to those from 6.5 years to 89 years of age.The test takes approximately 12-20 minutes to carry out and generates a number of psychometric scores, including numbers, percentages, and percentiles of: categories achieved, trials, errors, and perseverative errors. Can be interpreted as: the greater the percentage, the greater the measured ability.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Groups:
- Placebo/Control: Placebo/control
  Cognitive retraining : video
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
percentage of correct responses | 38.43 (24.07) | 35.79 (21.57) | 43.14 (27.06) | 39.57 (22.31)

2. Primary Outcome: Hopkins Verbal Learning Test
Description: The Hopkins Verbal Learning Test is designed to assess verbal learning and memory (immediate recall, delayed recall, delayed recognition). The assessment takes approximately 5-10 minutes with a 25-minute delay to complete and 2 minutes to score. The greater the score, the greater the measured recall. The score ranges from 0 to 24.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 20.74 (5.25) | 19.80 (5.94) | 20.42 (7.51) | 21.45 (5.85)

3. Primary Outcome: Spatial Span- Total Score
Description: The Spatial Span subtest of the Wechsler Memory Scale can be used as an indicator of working memory and visuospatial processing. An increase in severity of impairment results in a decrease in Spatial Span Total Score. The range is 1 to 28.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 13.59 (4.18) | 13.88 (4.20) | 13.21 (3.23) | 13.58 (4.07)

4. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: The PANSS is a handscored instrument. It uses 25 PANSS items organized into five scales: Negative, Positive, Dysphoric Mood, Activation, and Autistic Preoccupation. The PANSS is based on findings that schizophrenia comprises at least two distinct syndromes. The positive syndrome consists of productive symptoms, while the negative syndrome consists of deficit features. This distinction is useful when developing treatment plans because you can focus on the type of symptoms the patient is experiencing. It is also useful when studying the effects of medication (e.g., in clinical drug trials) because it allows you to determine which type of symptoms are being affected. PANSS Total score minimum = 30, maximum = 210. The greater the score, the greater the symptoms.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 53.30 (13.58) | 52.01 (13.34) | 53.79 (12.76) | 53.96 (12.43)

5. Secondary Outcome: Heinrichs-Carpenter Quality of Life Scale
Description: The Heinrichs-Carpenter Quality of Life Scale is a testing device. It has a range of possible scores, 0-126 used to evaluate social functioning & behavior in patients with schizophrenia-lower scores represent poorer mental health.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 67.26 (20.04) | 68.30 (25.59) | 63.25 (24.15) | 63.92 (19.53)

6. Secondary Outcome: Simpson-Angus Neurological Rating Scale
Description: Simpson-Angus Scale (SAS) is a 10-item rating scale that has been used widely for assessment in both clinical practice and research settings. Items are rated for severity on a 0-4 scale, with definitions given for each anchor point. The highest possible score is 40.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 1.41 (2.53) | 0.72 (1.73) | 1.04 (1.27) | 1.81 (2.25)

7. Secondary Outcome: UCSD Performance-Based Skills Assessment (UPSA)
Description: The UCSD Performance-Based Skills Assessment (UPSA) is a role-play test designed to evaluate a person's functional capacity in two selected areas of basic living skills. These areas include Finance and Communication. Subjects being tested utilize props to demonstrate how they perform everyday activities and are assessed on their actual performance. The higher the score, the better the performance of an individual. The scores range from 0 to 100.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Number analyzed (Participants) | 27 | 27 | 24 | 26
units on a scale | 34.19 (9.41) | 32.80 (10.98) | 32.60 (13.82) | 31.39 (10.01)

ADVERSE EVENTS:
Time Frame: Adverse events (serious and other) are reported overall at the month time frame.
Arm/Group | D-serine/Control | Placebo/Cog Rehab | D-serine/Cog Rehab | Placebo/Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/24 | 0/26
Other Adverse Events (participants affected / at risk) | 14/27 | 14/27 | 12/24 | 18/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | D-serine/Control (N=27) | Placebo/Cog Rehab (N=27) | D-serine/Cog Rehab (N=24) | Placebo/Control (N=26)
Concentration Difficulty (Psychiatric disorders) | 2 (2) | 2 (2) | 2 (2) | 3 (3)
Increased Fatigue (Psychiatric disorders) | 4 (5) | 3 (3) | 1 (1) | 4 (4)
Sleepiness (Psychiatric disorders) | 6 (15) | 7 (8) | 6 (12) | 9 (20)
Failed Memory (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (3) | 4 (4)
Depression (Psychiatric disorders) | 3 (3) | 2 (4) | 1 (2) | 3 (7)
Tension (Psychiatric disorders) | 2 (2) | 3 (3) | 2 (4) | 3 (6)
Increased Sleep (Psychiatric disorders) | 8 (13) | 5 (6) | 3 (6) | 6 (9)
Reduced Sleep (Psychiatric disorders) | 2 (2) | 2 (3) | 3 (4) | 1 (1)
Increased Dreams (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0) | 4 (5)
Emotional Indifference (Psychiatric disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (2)
Dystonia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rigidity (Nervous system disorders) | 4 (8) | 0 (0) | 3 (4) | 7 (12)
Hypokinesia (Nervous system disorders) | 2 (5) | 1 (1) | 1 (1) | 2 (5)
Hyperkinesia (Nervous system disorders) | 5 (11) | 1 (5) | 2 (4) | 5 (10)
Tremor (Nervous system disorders) | 2 (2) | 5 (6) | 3 (5) | 5 (14)
Akathesia (Nervous system disorders) | 2 (3) | 2 (3) | 2 (3) | 3 (6)
Epileptic Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesias (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Accommodation Distance (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased Salivation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Reduced Salivation (Gastrointestinal disorders) | 1 (1) | 1 (3) | 1 (1) | 2 (5)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (3) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (2)
Micturition Distance (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polyuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
Dizziness (General disorders) | 0 (0) | 2 (3) | 2 (3) | 4 (6)
Polyps / Tachycardia (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Increased Sweat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (5)
Increased Pigmentation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight Increase (Metabolism and nutrition disorders) | 2 (2) | 4 (6) | 3 (5) | 8 (12)
Weight Decrease (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 3 (8) | 2 (20) | 1 (3) | 0 (0)
Galactorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased Sexual Desire (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diminished Sexual Desire (Reproductive system and breast disorders) | 3 (5) | 1 (2) | 0 (0) | 2 (8)
Sexual Dysfunction (Reproductive system and breast disorders) | 3 (5) | 0 (0) | 0 (0) | 3 (11)
Tension Headache (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Migraine Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Physical Dependence (General disorders) | 2 (4) | 1 (4) | 0 (0) | 3 (5)
Psychological Dependence (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Other Headache (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No